CLINICAL TRIAL: NCT04913155
Title: HANSE - Holistic Implementation Study Assessing a Northern German Interdisciplinary Lung Cancer Screening Effort, Population-based Screening Study -Prospective, Randomized Comparator Controlled
Brief Title: HANSE - Holistic Implementation Study Assessing a Northern German Interdisciplinary Lung Cancer Screening Effort
Acronym: HANSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: LungenClinic Grosshansdorf (Other); University Hospital Schleswig-Holstein (Other); German Center for Lung Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ESR-20-20770
Record Dates: First submitted 2021-05-10; First posted 2021-06-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Screening program; Low-dose CT
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Population-based Screening Study -Prospective, randomized comparator controlled
Who Masked: Participant
Masking Description: Randomized reporting of coronary calcium score and emphysema score
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Reporting group (coronary calcium score and emphysema score) (Other): Coronary calcium score and emphysema score are reported to subjects
  Interventions: Radiation: Low-dose CT screening
- Reporting group (coronary calcium score only) (Other): Only coronary calcium score is reported to subjects
  Interventions: Radiation: Low-dose CT screening
- Reporting group (emphysema score only) (Other): Only emphysema score is reported to subjects
  Interventions: Radiation: Low-dose CT screening
- Non-reporting group (Other): Coronary calcium score and emphysema score are not reported to subjects
  Interventions: Radiation: Low-dose CT screening
- Low-risk group (No Intervention): No CT screening, collection of health data only

INTERVENTIONS:
Radiation: Low-dose CT screening — Low-dose computed tomography with lung nodule evaluation (LungRADS1.1, highrisk score group), randomized reporting of coronary artery calcium score and emphysema score
  Arms: Non-reporting group; Reporting group (coronary calcium score and emphysema score); Reporting group (coronary calcium score only); Reporting group (emphysema score only)

SUMMARY:
The HANSE study is primarily intended as a pilot to provide evidence that a holistic and effective lung cancer screening program can be implemented in Germany and that such a screening program can be integrated in the current infrastructure of certified lung cancer centers.

DETAILED DESCRIPTION:
Germany has a long history of offering screening programs for cancers, such as breast, colorectal, and, more recently, cervical and skin cancer. Screening for lung cancer, however, which causes more deaths than any other cancer in men and is the second leading cancer death in women (not far behind breast cancer), has not been implemented to date. Only very recently, Institute for Quality and Efficiency in Healthcare (IQWiG) in a preliminary assessment of low-dose CT screening, concluded that the benefits from screening outweigh potential risks. However, an implementation of a national lung cancer screening program, which would be covered by the general health insurance, will likely not be implemented before 2022.

Nonetheless, the IQWiG report also comments on important criteria for implementing lung cancer screening in Germany using low-dose CT:

1. It would be necessary to determine criteria that define a high-risk population. Various risk forecasting models are currently being propagated to enable a more precise selection of high-risk individuals. Their reliability and repeatability needs to be checked.
2. Integration of access to a smoking cessation program.
3. Quality assurance measures must be taken into account, including standardized protocols for the evaluation of the CT images and the subsequent follow-up checks as well as the invasive diagnostic tissue sampling procedures. The HANSE study is primarily intended as a pilot to provide evidence that a holistic and effective lung cancer screening program can be implemented in Germany and that such a screening program can be integrated in the current infrastructure of certified lung cancer centers.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 55-79 years
2. Current or former smokers
3. Subjects with calculated risk score PLCOM2012 ≥1.58% (6 yrs.) or NELSON inclusion criteria (current or former smokers [those who had quit ≤10 years ago] who had smoked >15 cigarettes a day for >25 years or >10 cigarettes a day for >30 years).
4. Able and willing to give written informed consent In addition, non-qualifying subjects fulfilling inclusion criteria 1 (age), 2 (smoking history) and 4 (consent), but do not meet the inclusion criterion 3 (risk too low) will be asked to volunteer by contributing long-term outcome data informing of the development of lung cancer or death from lung cancer (about n=7100 randomly selected from all 3 centers, low-risk group). These subjects will be contacted via mail after a minimum of 5 year follow up to inquire if they developed lung cancer in the time between their recruitment and present. Non-responders will be followed by local registries and by phone. New lung cancer cases will be verified using official hospital or cancer registry documents.

Exclusion Criteria:

1. Comorbidity, which would unequivocally contraindicate either screening or treatment if lung cancer is detected.
2. History of chest CT within the past year preceding the invitation.
3. Inability to undergo non-contrast CT (e.g. ≥ 200 kg body weight, inability to lie flat).
4. Pregnancy
5. Risk of non-compliance with study procedures.

   * Unable to give written consent
   * Patient's inability to fill in the questionnaire self-dependent
   * Limited knowledge of the German language
   * Inability to travel, residents of care facilities, etc.

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12100 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 5 years
  Positive predictive value (PPV) for lung cancer detection with different inclusion methods (NELSON vs. PLCO) after 2 screening rounds.

SECONDARY OUTCOMES:
Key secondary endpoint 1 | 1 year
  Proportion of individuals selected for screening within the high-risk population.
Key secondary endpoint 2 | 5 years
  Proportion of lung cancers detected with different inclusion methods (NELSON vs. PLCO) within the overall study population after 5 years.
Key secondary endpoint 3 | 5 years
  Proportion of lung cancers detected with in the high-risk population after 5 years.
Key secondary endpoint 4 | 5 years
  Specificity within the overall population after 5-year follow-up.
Key secondary endpoint 5 | 5 years
  Sensitivity within the overall population after 5-year follow-up.
Additional secondary endpoint 1 | 1 year
  Rate of initiation of cardiovascular treatments (in particular lipid-lowering) in the calcium score reporting group vs. the non-reporting group after year 1 of study.
Additional secondary endpoint 2 | 1 year
  Efficiency of nodule management algorithms (LungRads1.1 + PanCan) will be evaluated according to the number of patients sorted in the category (a) "Next surveillance scan" AND the number of patients with lung cancer sorted into category (b) "early recall scan", or (c) "diagnostic evaluation".
Additional secondary endpoint 3.1 | 1 year
  Success of screening program. Based on all individuals enrolled. Definition of success is calculated using Response rate.
Additional secondary endpoint 3.2 | 1 year
  Success of screening program. Based on all individuals enrolled. Definition of success is calculated using Reliability of PLCO risk scoring (self-reported vs. on site assessment).
Additional secondary endpoint 3.3 | 1 year
  Success of screening program. Based on all individuals enrolled. Definition of success is calculated using Percentage of subjects receiving an adequate low-dose CT scan and report according to DRG guidelines (number of diagnostic CTs/number of all CTs).
Additional secondary endpoint 3.4 | 1 year
  Success of screening program. Based on all individuals enrolled. Definition of success is calculated using Percentage of subjects receiving adequate follow-up procedures.
Additional secondary endpoint 4.1 | 1 year
  Quality of screening program: CT reading performance (2nd reader vs. CAD vs. AI)
Additional secondary endpoint 4.2 | 1 year
  Quality of screening program: Quality of lung nodule management
Additional secondary endpoint 4.3 | 1 year
  Quality of screening program: Frequency of detection and management of incidental findings from low dose chest CT (emphysema, coronary heart disease, etc.)
Additional secondary endpoint 4.4 | 1 year
  Quality of screening program: LDCT dose management
Additional secondary endpoint 5 | 1 year
  Smoking cessation: Success of smoking cessation counseling based on number of participants quitting with or without revealing additional health risks (emphysema score, coronary calcium score or both).
Additional secondary endpoint 6.1 | 1 year
  Identification of blood-based biomarkers for early detection of lung tumors: Blood collection and evaluation of various blood-based epigenetic biomarkers in positive LDCT cases with subsequent biopsy on the positive predictive value of the LDCT test.
Additional secondary endpoint 6.2 | 1 year
  Identification of exhalation-based biomarkers for early detection of lung tumors: Collection of breath condensate and evaluation of various exhalation-based epigenetic biomarkers in positive LDCT cases with subsequent biopsy on the positive predictive value of the LDCT test.
Additional secondary endpoint 7.1 | 1 year
  Cost-effectiveness analysis: Main objectives of the modelling study are to investigate the impact of different components of LDCT lung cancer screening on the long-term all-cause mortality and cost-effectiveness. Key components include risk score-based selection criteria, nodule management protocols, threshold values of imaging biomarkers for cardio-vascular diseases and COPD, and inclusion of smoking cessation programs (performed by Center for Health Economics Research Hannover (CHERH).
Additional secondary endpoint 7.2 | 1 year
  Cost-effectiveness analysis: Comparison of patient recruitment strategies: Cost-effectiveness of register-based mailing campaign vs. GP referrals in terms of recruitment of qualified screening subjects (Center for Health Economics Research Hannover - CHERH).

CONTACTS AND LOCATIONS:
Overall Officials: Jens Vogel-Claussen, Prof. Dr., Study Director — Hannover Medical School
Locations (3):
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - LungenClinic Grosshansdorf, Großhansdorf, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogel-Claussen J, Bollmann BA, May K, Stiebeler S, Dettmer S, Faron A, Kuhlmann A, Schmid-Bindert G, Kaaks R, Barkhausen J, Bohnet S, Reck M; HANSE investigators. Effectiveness of NELSON versus PLCOm2012 lung cancer screening eligibility criteria in Germany (HANSE): a prospective cohort study. Lancet Oncol. 2025 Dec;26(12):1541-1551. doi: 10.1016/S1470-2045(25)00490-5. Epub 2025 Nov 10. PMID 41232542
- See also: Study web page (German language) — https://www.hanse-lungencheck.de

DOCUMENTS (2):
  • Study Protocol: Study amendment (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT04913155/Prot_000.pdf
  • Study Protocol: Main protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT04913155/Prot_001.pdf